CLINICAL TRIAL: NCT00860535
Title: A Multicenter Phase Ib Trial to Determine Whether a Gene Expression Signature Changes in Response to Treatment With Bcr-Abl Inhibitors in Patients With Blast Phase Philadelphia Chromosome Positive Chronic Myelogenous Leukemia or Philadelphia Chromosome Positive Acute Lymphocytic Leukemia
Brief Title: Growth Factor Signature (GFS) Pilot Study (MK0000-098)(COMPLETED)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0000-098; 2009_558
Record Dates: First submitted 2009-03-05; First posted 2009-03-12 (Estimated); Results first posted 2011-10-10 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Blast Phase Philadelphia Chromosomes Positive (Ph+) Chronic Myelogenous Leukemia (CML); Philadelphia Chromosome Positive (Ph+) Acute Lymphocytic Leukemia (ALL)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ph+ CML or Ph+ ALL (Experimental): GFS biomarker evaluation
  Interventions: Other: Comparator: Biomarker evaluation

INTERVENTIONS:
Other: Comparator: Biomarker evaluation — Patients on standard of care treatment will have blood drawn to evaluate biomarker changes in response to treatment with BCR-ABL inhibitors over a ~3.5 month period.
  Part I will enroll patients who are beginning treatment with imatinib (recommended dose 400 mg every day [qd]), dasatinib (recommended dose 70 mg twice a day [bid]), or nilotinib (recommended dose 400 mg bid).
  Part II will enroll patients who are changing from imatinib therapy to either dasatinib or nilotinib. A decision to initiate Part II will be made based on analysis of the results of Part I.

SUMMARY:
This study will evaluate a gene expression signature (Growth Factor Signature [GFS]) as a biomarker for response/resistance to BRC-ABL oncogene inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a histologically or cytopathologically confirmed blast phase Ph+ CML or Ph+ ALL.
* Participant is 18 years of age on the day of signing informed consent
* Participant must have performance status 0-3 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Participant has at least 30 percent blasts in peripheral blood; or at least 30 percent lymphoblasts in peripheral blood or bone marrow

  * For Part II:
* Participant has progressed while taking imatinib or is unable to tolerate imatinib, being defined as discontinuing imatinib treatment as a result of nonhematologic toxic effects of any grade
* If female, participant is either post-menopausal, free from menses for >2 years, surgically sterilized or willing to use 2 adequate barrier methods of contraception to prevent pregnancy or agrees to abstain from heterosexual activity throughout the study, starting with Visit 1
* Female participants of childbearing potential must have a negative serum or urine pregnancy test (beta hCG) at screening
* If male, participant is surgically sterilized, agrees to use an adequate method of contraception, or agrees to abstain from heterosexual activity for the duration of the study
* Participant or the patrticipant's legal representative has voluntarily agreed to participate by giving written informed consent
* Participant must be available for periodic blood sampling, study related assessments, and management at the treating institution for the duration of the study

Exclusion Criteria:

* Participant is currently participating in or has participated in a study with an investigational compound or device within 30 days or 5 half-lives, whichever is longer, of the start of treatment
* Participant has known human immunodeficiency virus (HIV) infection or HIV-related malignancy
* Participant is a female who is pregnant or breastfeeding, or is expecting to conceive within the projected duration of the study
* Participant has a known allergy or hypersensitivity to imatinib, dasatinib or nilotinib
* Participant has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate
* Participant has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* There is any concern by the investigator regarding the safe participation of the participant in the study or for any other reason, the investigator considers the participant inappropriate for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Ph+ CML or Ph+ ALL: Participants with blast phase Philadelphia Chromosomes Positive (Ph+) Chronic Myelogenous Leukemia (CML) or Philadelphia Chromosome Positive (Ph+) Acute Lymphocytic Leukemia (ALL) who were beginning treatment with imatinib, dasatinib or nilotinib as per standard of care. All participants who had evaluable gene expression data were included in the analysis.
Period: Overall Study
Arm/Group | Ph+ CML or Ph+ ALL
Started | 9
DISCONTINUED | 1 (Participant did not meet inclusion criteria and did not complete the study.)
Completed | 8
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Ph+ CML or Ph+ ALL: Growth Factor Signature (GFS) biomarker evaluation in participants with blast phase Ph+ CML or Ph+ ALL who were treated with imatinib, dasatinib or nilotinib as per standard of care.
Arm/Group | Ph+ CML or Ph+ ALL
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Growth Factor Signature (GFS) Variability at Baseline
Description: The GFS was measured by microarray analysis using the entire 101 gene signature. The GFS is quantified as the change in gene expression between two separate samples collected from the same patient. The signature has 101 genes in two oppositely regulated arms, which are pre-specified. The expression of genes in the UP arm goes up with increasing pathway activity, and the expression of genes in the DOWN arm goes down with increasing pathway activity.
  The GFS variability was represented by the GFS change between two baseline samples (Mean GFS Fold Ratio [Screening to Day 1 Predose]).
Time Frame: Screening to Day 1 Predose
Population: Participants whose GFS was measured using microarrays to determine the pretreatment baseline variability in participants with blast phase Ph+ CML or Ph+ ALL.
Measure: Mean (90% Confidence Interval); unit: GFS Fold Ratio-Screening to Day1 Predose
Groups:
- Ph+ CML or Ph+ ALL: Participants with blast phase Ph+ CML or Ph+ ALL who were beginning treatment with imatinib, dasatinib or nilotinib as per standard of care. All participants who had evaluable gene expression data were included in the analysis.
Arm/Group | Ph+ CML or Ph+ ALL
Number analyzed (Participants) | 8
GFS Fold Ratio-Screening to Day1 Predose | 1.11 (0.90) [1.03 to 1.21]

2. Primary Outcome: Growth Factor Signature (GFS) Change From Baseline Measured by Time Weighted Average (TWA) for Days 1 to 22
Description: The GFS was measured by microarray analysis using the entire 101 gene signature.
  The TWA is the area under the curve (AUC) divided by the time interval (for this study it was the AUC of gene-expression divided by Days 1 to 22).
  Participants with blast phase Ph+ CML or Ph+ ALL were measured for change in the GFS post-treatment when treated with imatinib, dasatinib, or nilotinib, using Microarray. Change was represented as the GFS Fold Ratio of TWA for Days 1 to 22 to Baseline.
Time Frame: Baseline to 22 Days After Initiation of Therapy
Measure: Mean (90% Confidence Interval); unit: GFS Fold Ratio-TWA[Days1-22] to baseline
Arm/Group | Ph+ CML or Ph+ ALL
Number analyzed (Participants) | 9
GFS Fold Ratio-TWA[Days1-22] to baseline | 0.74 [0.66 to 0.83]

ADVERSE EVENTS:
Time Frame: All participants in the study were followed for all clinical adverse experiences from baseline until 5 days following any protocol specific procedure.
Groups:
- Ph+ CML or Ph+ ALL: Participants with blast phase Ph+ CML or Ph+ ALL who were beginning treatment with imatinib, dasatinib or nilotinib as per standard of care.
Arm/Group | Ph+ CML or Ph+ ALL
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Part I aimed to have 10 evaluable patients. Due to slow enrollment, 9 patients who met the inclusion/exclusion criteria were enrolled over a period of 9 months. Part I was terminated early and Part II was cancelled due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No